CLINICAL TRIAL: NCT00983138
Title: Efficacy and Safety of Recombinant Asparaginase in Infants (<1 Year) With Previously Untreated Acute Lymphoblastic Leukaemia - Phase II Clinical Trial
Brief Title: Efficacy and Safety of Recombinant Asparaginase in Infants With Previously Untreated Acute Lymphoid Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Cécile Guimbal-Schmolck, PhD, medac GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-ASP.6/INF; EudraCT No: 2008-006300-27
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Acute Lymphoid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recombinant asparaginase (Experimental)
  Interventions: Drug: recombinant asparaginase

INTERVENTIONS:
Drug: recombinant asparaginase — 10 000 Units/m² adjusted to age, 6 i.v. infusions (day 15, day 18, day 22, day 25, day 29, day 33) during the induction therapy

SUMMARY:
This non-controlled multicentre phase II study is designed to assess the safety and to describe (in relation to children of higher age) the pharmacodynamics of recombinant ASNase (rASNase) for first-line treatment of infants (< 1 year of age at diagnosis) with de novo acute lymphoblastic leukaemia

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated T-lineage or precursor B-lineage ALL or biphenotypic leukaemia according to EGIL criteria.
* Morphological verification of the diagnosis, confirmed with cyto¬chemistry and immunophenotyping.
* Age < 1 year at diagnosis.
* Written informed consent of the parents or other legally authorised guardian of the patient.
* Treatment according to protocol INTERFANT 06

Exclusion Criteria:

* Mature B-lineage ALL, defined by the immunophenotypical presence of surface immunoglobulins or t(8;14) and breakpoint as in B-ALL.
* The presence of the t(9;22)(q34;q11) or bcr-abl fusion in the leukaemic cells.
* Systemic use of corticosteroids less than 4 weeks before diagnosis. Patients who received corticosteroids by aerosol are eligible.
* Known allergy to any ASNase preparation.
* Pre-existing known coagulopathy (e.g. haemophilia).
* Pre-existing pancreatitis.
* Liver insufficiency (bilirubin > 50 µmol/L; SGOT/SGPT > 10 x the upper limit of normal).

Max Age: 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
number of patients with hypersensitivity reactions to rASNase | within 2 months

SECONDARY OUTCOMES:
pharmacodynamic of rASNase | within 33 days

CONTACTS AND LOCATIONS:
Overall Officials: Rob Pieters, MD, Principal Investigator — Erasmus MC-Sophia Children's Hospital
Locations (17):
- Germany (11):
  - Hospital Charité Virchow, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - University Hospital Johann Wolfgang Goethe, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Medical University Hannover, Hanover
  - University Hospital Schleswig-Holstein, Campus Kiel, Kiel
  - University Hospital Münster, Münster
  - Olga Hospital, Stuttgart
- Netherlands (6):
  - VU University Medical Centre, Amsterdam
  - Academic Medical Centre AMC/EK2, Amsterdam
  - University of Groningen, Groningen
  - University Children's Hospital Nijmegen, Nijmegen
  - Sophia Children's Hospital, Rotterdam
  - University Medical Centre Utrecht, Utrecht